CLINICAL TRIAL: NCT04820166
Title: The Effect of Monitoring Portal Venous Pressure on Clinical Outcomes in Patients With Portal Hypertension: a Prospective, Single-center, Observational Study
Brief Title: The Effect of Monitoring PVP on Clinical Outcomes in Patients With PH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-062
Record Dates: First submitted 2021-03-18; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: monitoring portal pressure gradient or hepatic venous pressure gradient — measuring portal pressure gradient or hepatic venous pressure gradient regularly

SUMMARY:
The complications associated with portal hypertension in cirrhosis are the main cause of death in patients with cirrhosis. The level of portal venous pressure is closely related to the prognosis of patients. HVPG (hepatic venous pressure gradient) is the "gold standard" for predicting portal venous pressure and an important indicator for evaluating the efficacy of NSBBS. However, monitoring HVPG has many limitations，and the clinical application is also limited to a certain extent. Therefore, this study intends to clarify the guiding value of monitoring portal venous pressure in the clinical diagnosis and treatment of portal hypertension patients through a single-center, prospective and observational study. Therefore, this study intends to clarify the guiding value of monitoring portal venous pressure in the clinical diagnosis and treatment of portal hypertension patients through a single-center, prospective and observational study. At the same time, to explore the correlation between HVPG and PPG in cirrhosis patients at different stages and different etiologies, and to evaluate the role of spleen stiffness in predicting the severity of esophageal and gastric varices in patients with portal hypertension, and to find biomarkers to predict the risk of complications related to portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* With chronic liver disease
* Age 18-80 years
* Patients who require a portal pressure measurement at the discretion of the treating physician
* Voluntarily signed informed consent

Exclusion Criteria:

* With serious cardiopulmonary disease or other diseases affect survival
* With severe renal dysfunction
* Concomitant portal vein cavernous degeneration or extensive portal vein thrombosis
* Women who are planning to become pregnant or who are pregnant or breastfeeding
* The researcher judged that it was not suitable to participate in this study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with portal hypertension
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastroesophageal varices bleeding | three years
  Patients with gastroesophageal varices has hematemesis or melena, and active bleeding or red sign can be seen under endoscopy
Ascites | three years
  Peritoneal effusion was seen under ultrasound
Hepatic encephalopathy | three years
  Patients with altered consciousness or unresponsiveness, accompanied by elevated blood ammonia

SECONDARY OUTCOMES:
Death or final follow-up time (3 years) | three years

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu M, Zhang X, Cheng X, He Q, Zhou T, Wang H, Li B, Luo W, Li J, Li H, Lin Z, Song J, Wang W, Huang J, Ji Y, Zhou D, Xie W, Yang Q, Tu M, Luo X, Zhang X, Yan H, Chen J. Indocyanine Green Clearance Test via Pulse Dye Densitometry for Portal Hypertension Diagnosis in cACLD. Liver Int. 2025 Dec;45(12):e70425. doi: 10.1111/liv.70425. PMID 41178521
- [Derived] Zhang X, Zhou L, Liang W, Cheng X, He Q, Li H, Luo W, Huang J, Li J, Wang W, Tu M, Wang H, Ou P, Wen B, Xiao L, Zhou D, Wong VW, Chen J. Identification of Clinically Significant Portal Hypertension in cACLD Individuals With Spleen Stiffness Measurement. Liver Int. 2025 Apr;45(4):e16241. doi: 10.1111/liv.16241. PMID 40105356